CLINICAL TRIAL: NCT01600144
Title: Data Collection for CAD Evaluation
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s53792
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Data Collection
Keywords: data mammography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- data collection
  Interventions: Other: digital mammography

INTERVENTIONS:
Other: digital mammography — data collection

SUMMARY:
Mammographical data collection (raw data) for CAD evaluation by VUCOMp software.

ELIGIBILITY:
Inclusion Criteria:

* women who underwent a digital mammography imaging

Exclusion Criteria:

* men

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: women
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-03 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Datacollection | 2 years
  No outcome described, only datacollection

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Van Ongeval, MR,Phd, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Belgium